CLINICAL TRIAL: NCT01061645
Title: Phase I Study of MOC31-PE in Antigen Positive Carcinomas
Brief Title: Study of MOC31-PE in Antigen Positive Carcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, Senior Physician, Oslo University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOC31-PE
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Carcinoma
Keywords: MDT and DLT
MeSH Terms: conditions — Carcinoma; Anemia, Dyserythropoietic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MOC31-PE (Experimental)
  Interventions: Drug: MOC31-PE

INTERVENTIONS:
Drug: MOC31-PE — Immunotoxines

SUMMARY:
Immunotoxins (ITs), monoclonal antibodies conjugated to plant or bacterial toxins, have been extensively investigated for their possible use as anti-tumor agents although not in carcinoma patients with minimal residual disease. Various ITs have been tested in early clinical trials and recent studies demonstrate anti-tumor activity of IT treatment in patients with glioblastoma and different solid tumors. Systemic treatment with immunotoxins directed against carefully selected epithelial cell surface molecules may have a potential for eradicating also dormant metastatic tumor cells, as their action is independent of cell proliferation. The effector moieties of the IT used here, the Pseudomonas exotoxin A (PE), inhibits protein synthesis in eukaryotic cells by catalytic inactivation (ribosylation) of elongation factor 2 in the ribosome complex.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirm epithelial carcinoma, verified to be positive for the targeting antigen(Ep-CAM/epithelial glyco protein 2)according to the criteria given below.
* Tumor specimens verified to be positive for the targeting antibody,i.e.EGP2 positive (MOC31) by immunocytochemical or histochemical staining.
* Signed written informed consent
* Patients with no clinically symptomatic central nervous system (CNS) involvement.
* Both gender, age 18 -75 years old.
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Adequate hematologic, renal and hepatic function defined as: Neutrophils > 1.5 x 10^9/L;Platelets > 100 x 10^9/L; Creatinine < 120 umol/L; Total bilirubin within normal range. Liver enzymes (ALAT and ASAT <2.5 UNL: alkaline phosphatase < 1.5 UNL and yGT < 1.5 UNL).
* Coagulation parameters (pT, PTT) within normal range.

Exclusion Criteria:

* No medical history of Hepatitis B or C infection
* Patients must have no ECG abnormalities
* Patients must not be HIV positive
* Female premenopausal patients should not be pregnant (must have a negative pregnancy test prior to inclusion) and should not be lactating.
* Patients must use effective contraception if of reproductive potential.
* Prior chemotherapy and/or radiation should be completed for at least 4 weeks prior to study enrolment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The documentation of the Maximum Tolerated Dose (MID) | 2 years
The identification of the dose limiting toxicity (DLT) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Norwegian Radium Hospital, Department of Clinical Cancer Research, Oslo, Norway